CLINICAL TRIAL: NCT05619861
Title: Clinical Study of CAR-T Technique in the Treatment of Recurrent and Refractory Hematopoietic and Lymphatic Tumor
Brief Title: CAR-T Cells in the Treatment of Malignant Hematological Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Collaborators: Cangzhou People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022/11/09
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Lymphoma, B-Cell; Leukemia, B-cell; Leukemia, T-Cell; Multiple Myeloma
Keywords: T cells
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, B-Cell; Leukemia, T-Cell; Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T (Experimental): Autologous CAR-T cells, intravenous infusion, infusion dose 0.1-3 × 106CAR-T cells/kg
  Interventions: Biological: CAR-T

INTERVENTIONS:
Biological: CAR-T — Patients will receive CAR-T treatment

SUMMARY:
To evaluate the safety of autologous CAR-T cell injection in the treatment of recurrent and refractory hematopoietic and lymphoid tissue tumors

DETAILED DESCRIPTION:
Main research objective: To evaluate the safety of autologous CAR-T cell injection in the treatment of recurrent and refractory hematopoietic and lymphoid tissue tumors. Secondary research objective: To investigate the efficacy and cytodynamic characteristics of autologous CAR-T cell injection in the treatment of recurrent and refractory hematopoietic and lymphoid tissue tumors

ELIGIBILITY:
1. With the consent of himself or the legal guardian and the signed informed consent, he is willing and able to comply with the planned visit, research and treatment, laboratory examination and other test procedures; Clinical Study of CAR-T Technique in the Treatment of Recurrent and Refractory Hematopoietic and Lymphatic Tumor
2. Patients with recurrent and refractory hematopoiesis and lymphoid tissue tumors determined by clinical diagnosis;
3. Age 14-70 (including boundary value), both male and female;
4. Subjects with a physical status of 0~2 in the American Eastern Oncology Collaboration Group (ECOG);
5. The results of treatment related antigens were positive;
6. The expected life span is more than 3 months from the date of signing the informed consent;

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-04-27 (Actual); Primary Completion 2023-01-26 (Estimated); Study Completion 2023-12-26 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence and severity of adverse events | 24 months post CAR-T cells infusion
  The incidence and severity of adverse events and adverse reactions from infusion to withdrawal or before the safety follow-up period

CONTACTS AND LOCATIONS:
Locations (1):
- Cangzhou People's Hospital, Cangzhou, Hebei, China